CLINICAL TRIAL: NCT06740188
Title: Impact of Trazodone on Non-rapid Eye Movement Sleep Stage Ⅲ in Depressed Insomniac Co-morbid Patients: a Randomized Controlled Trial
Brief Title: Trazodone on NREM Sleep Stage Ⅲ in Depressed Insomniac Co-morbid Patients
Acronym: n-REMSS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jie Tong, Prof., Tongji University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PWRq2024-21
Record Dates: First submitted 2024-12-11; First posted 2024-12-18 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-12

CONDITIONS: Depressed Insomniac Co-morbid Patients
Keywords: Trazodone; Non-rapid Eye Movement Sleep Stage; depression; insomnia
MeSH Terms: conditions — Depression; Sleep Initiation and Maintenance Disorders | interventions — Zolpidem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group was given only 5-hydroxytryptamine balanced antidepressants trazodone.
  Interventions: Drug: 5-hydroxytryptamine balanced antidepressants trazodone
- Control group (Active Comparator): The control group was given citalopram hydrobromide combined with zolpidem.
  Interventions: Drug: Citalopram hydrobromide combined with zolpidem

INTERVENTIONS:
Drug: 5-hydroxytryptamine balanced antidepressants trazodone — The intervention group was given only 5-hydroxytryptamine balanced antidepressants trazodone
  Arms: Intervention group
Drug: Citalopram hydrobromide combined with zolpidem — the control group was given citalopram hydrobromide combined with zolpidem
  Arms: Control group

SUMMARY:
This study used polysomnographic technology and randomly selected 60 patients who met the diagnostic criteria for depression and non-organic insomnia as stipulated in DSM-5 into an intervention group (n=30) and a control group (n=30). The intervention group was given only 5-hydroxytryptamine balanced antidepressants trazodone, while the control group was given citalopram hydrobromide combined with zolpidem. Both groups underwent PSG at baseline and 1 week after medication, and were assessed with the 17-item Hamilton Depression Rating Scale, Zung Self-Rating Depression Scale, Pittsburgh Sleep Quality Index, Arnsworth Insomnia Severity Scale, Antidepressant Side Effects Checklist, and the Drug Dependence Scale neuropsychological assessment at baseline, 1, 2, and 4 weeks after medication. The study aimed to explore the effects of single use of SMAs class antidepressants versus combination with other antidepressants on non-rapid eye movement sleep stage III in patients with depression and insomnia comorbidity, and to compare the effects of depression and insomnia in the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Outpatient or inpatient patients;
* 18 years old ≤ 65 years old;
* Simultaneously meet the diagnostic criteria for depression and non organic insomnia in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) in the United States;
* 17 items of Hamilton Depression Rating Scale (HAMD-17) with a total score of ≥ 17 points;
* Pittsburgh Sleep Quality Index (PSQI) ≥ 16 points;
* Never used related antidepressants and sedative hypnotic drugs;
* Has a certain level of visual and auditory resolution, and no comprehension barriers;
* Capable of independently completing scale measurements;
* Education level above primary school;
* Obtain written informed consent from the patient, and obtain written informed consent from the legal guardian if the patient is incapacitated during the onset of the illness.

Exclusion Criteria:

* Patients with comorbidities such as schizophrenia, schizophrenia, bipolar disorder, mental retardation, pervasive developmental disorder, delirium, dementia, cognitive impairment, alcohol dependence, etc
* Suffering from serious organic diseases, such as diabetes, thyroid disease, hypertension, cardiovascular disease, craniocerebral trauma, cerebral ischemia or hemorrhage;
* Patients with narrow angle glaucoma;
* History of epilepsy and febrile seizures;
* Individuals with a history of drug use;
* Positive for syphilis specific antibody and AIDS antibody;
* According to risk assessment, there are currently serious suicide attempts or individuals who are overly agitated Pregnant or lactating women, or those planning to conceive in the near future;
* Laboratory tests indicate the presence of liver and kidney function impairment in individuals;
* There are other individuals who meet the relevant contraindications for antidepressants.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep structure staging | Baseline and 1 week after medication
  Monitoring sleep structure staging through Polysomnography（PSG）:
  W period (awake period): Refers to the time when one has not entered a sleep state； N1 stage (non rapid eye movement stage 1): light sleep stage, accounting for about 5-10%； N2 stage (non rapid eye movement stage 2): The main part of sleep, accounting for about 50%； N3 stage (non rapid eye movement stage 3): Deep sleep stage, accounting for about 20%, is crucial for memory consolidation and recovery； R phase (rapid eye movement phase): related to dreams, accounting for about 20-25%.

SECONDARY OUTCOMES:
The 17 item Hamilton Depression Scale (HAMD-17) | baseline, 1, 2, and 4 weeks after medication
  The 17 item Hamilton Depression Scale (HAMD-17) evaluates the severity of depression and treatment outcomes in patients. Composed of 17 items, ranging from 7 to 13 points, it is classified as mild depression; 14-19 points are classified as moderate depression; ≥ 20 points is classified as severe or above.
Zong's Self rating Depression Scale (SDS) | baseline, 1, 2, and 4 weeks after medication
  Zong's Self rating Depression Scale (SDS): It can intuitively reflect the subjective feelings of depressed patients and their symptom changes during treatment. Composed of 20 items, the severity is rated on a 4-point scale from 1 to 4, with 53-62 indicating mild depression, 63-72 indicating moderate depression, and ≥ 72 indicating severe depression.
The Pittsburgh Sleep Quality Index (PSQI) | baseline, 1, 2, and 4 weeks after medication
  The Pittsburgh Sleep Quality Index (PSQI) evaluates a patient's sleep quality over the past month, including sleep outcomes and duration. There are a total of 18 items and 7 dimensions, each item is rated on a 4-point scale from 0 to 3. The higher the score, the worse the sleep quality.
The Athens Insomnia Scale (AIS) | baseline, 1, 2, and 4 weeks after medication
  The Athens Insomnia Scale (AIS) can be used as a subjective evaluation of insomnia in patients. Composed of 8 items, the severity is evaluated using a 4-point scale from 0 to 3, with a total score range of 0 to 24 points. The higher the score, the worse the sleep quality.
The Antidepressant Side Effect Checklist (ASEC) | baseline, 1, 2, and 4 weeks after medication
  The Antidepressant Side Effect Checklist (ASEC) evaluates the adverse reactions of patients after using antidepressants, including physical fatigue, dizziness, headache, sleep disturbances, erectile dysfunction, palpitations, tremors, sweating, dry mouth, constipation, urinary disorders, drowsiness, sexual dysfunction, and other symptoms. Composed of 21 items, the severity is evaluated using a 4-point scale from 0 to 3, with higher scores indicating more severe side effects. evaluates the adverse reactions of patients after using antidepressants, including physical fatigue, dizziness, headache, sleep disturbances, erectile dysfunction, palpitations, tremors, sweating, dry mouth, constipation, urinary disorders, drowsiness, sexual dysfunction, and other symptoms. Composed of 21 items, the severity is evaluated using a 4-point scale from 0 to 3, with higher scores indicating more severe side effects.
Drug Dependence Scale (DDS) | baseline, 1, 2, and 4 weeks after medication
  Drug Dependence Scale (DDS) used to identify the degree of drug use dependence. This scale adopts a 4-point rating system, with higher scores indicating higher levels of drug dependence.

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Geyer JD, Carney PR, Dillard SC, Davis L, Ward LC. Antidepressant medications, neuroleptics, and prominent eye movements during NREM sleep. J Clin Neurophysiol. 2009 Feb;26(1):39-44. doi: 10.1097/WNP.0b013e318196046f. PMID 19151617
- [Background] Sheehan DV, Rozova A, Gossen ER, Gibertini M. The efficacy and tolerability of once-daily controlled-release trazodone for depressed mood, anxiety, insomnia, and suicidality in major depressive disorder. Psychopharmacol Bull. 2009;42(4):5-22. PMID 20581790
- [Background] Sheehan DV, Croft HA, Gossen ER, Levitt RJ, Brulle C, Bouchard S, Rozova A. Extended-release Trazodone in Major Depressive Disorder: A Randomized, Double-blind, Placebo-controlled Study. Psychiatry (Edgmont). 2009 May;6(5):20-33. PMID 19724732
- [Background] Roth AJ, McCall WV, Liguori A. Cognitive, psychomotor and polysomnographic effects of trazodone in primary insomniacs. J Sleep Res. 2011 Dec;20(4):552-8. doi: 10.1111/j.1365-2869.2011.00928.x. Epub 2011 May 30. PMID 21623982
- [Background] Jarema M, Dudek D, Landowski J, Heitzman J, Rabe-Jablonska J, Rybakowski J. [Trazodon--the antidepressant: mechanism of action and its position in the treatment of depression]. Psychiatr Pol. 2011 Jul-Aug;45(4):611-25. Polish. PMID 22232986
- [Background] Collins PY, Patel V, Joestl SS, March D, Insel TR, Daar AS; Scientific Advisory Board and the Executive Committee of the Grand Challenges on Global Mental Health; Anderson W, Dhansay MA, Phillips A, Shurin S, Walport M, Ewart W, Savill SJ, Bordin IA, Costello EJ, Durkin M, Fairburn C, Glass RI, Hall W, Huang Y, Hyman SE, Jamison K, Kaaya S, Kapur S, Kleinman A, Ogunniyi A, Otero-Ojeda A, Poo MM, Ravindranath V, Sahakian BJ, Saxena S, Singer PA, Stein DJ. Grand challenges in global mental health. Nature. 2011 Jul 6;475(7354):27-30. doi: 10.1038/475027a. No abstract available. PMID 21734685